CLINICAL TRIAL: NCT06102395
Title: EFFECT-neo: A Prospective, Open-label, Multicenter Phase III Study to Evaluate Efficacy and Safety of Pembrolizumab Combined With Standard Chemotherapy in the Neoadjuvant Treatment of Local Advanced (LA) HNSCC
Brief Title: Evaluating the Efficacy and Safety of Pembrolizumab Plus Standard Chemotherapy in the Neoadjuvant Treatment of Local Advanced (LA) HNSCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT23456
Record Dates: First submitted 2023-04-12; First posted 2023-10-26 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Neoadjuvant Therapy; Pembrolizumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Cisplatin; Carboplatin; nedaplatin; Taxes; Docetaxel; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab combined with standard chemotherapy (Experimental): Patients receive pembrolizumab 200mg, IV, on day1 of Q3W; plus platinum (cisplatin 75 mg/m^2, IV, day 1 of Q3W or carboplatin AUC (area under curve) 2, IV, day 1-3 of Q3W or nedaplatin 80-100 mg/m^2, IV, day 2-4 of Q3W); plus other chemotherapy（nab-paclitaxel 260 mg/m^2, IV, day 1 of Q3W or docetaxel 75 mg/m^2, IV, day 1 of Q3W or liposomal paclitaxel 135-175 mg/m^2, IV, day 1 of Q3W or fluorouracil 750 mg/m^2, IV, day 1-5 of Q3W）; total 2 cycle
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Nedaplatin; Drug: Nab paclitaxel; Drug: Docetaxel; Drug: Liposomal paclitaxel; Drug: Fluorouracil
- Standard chemotherapy (Active Comparator): Patients receive platinum (cisplatin 75 mg/m^2, IV, day 1 of Q3W or carboplatin AUC (area under curve) 2, IV, day 1-3 of Q3W or nedaplatin 80-100 mg/m^2, IV, day 2-4 of Q3W); plus other chemotherapy（nab-paclitaxel 260 mg/m^2, IV, day 1 of Q3W or docetaxel 75 mg/m^2, IV, day 1 of Q3W or liposomal paclitaxel 135-175 mg/m^2, IV, day 1 of Q3W or fluorouracil 750 mg/m^2, IV, day 1-5 of Q3W）; total 2 cycle
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Nedaplatin; Drug: Nab paclitaxel; Drug: Docetaxel; Drug: Liposomal paclitaxel; Drug: Fluorouracil

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg, IV, on day1 of Q3W, 2 cycle
  Arms: Pembrolizumab combined with standard chemotherapy
Drug: Cisplatin — Cisplatin 75 mg/m^2, IV, day 1 of Q3W
Drug: Carboplatin — Carboplatin AUC (area under curve) 2, IV, day 1-3 of Q3W
Drug: Nedaplatin — Nedaplatin 80-100 mg/m^2, IV, day 2-4 of Q3W
Drug: Nab paclitaxel — Nab paclitaxel 260 mg/m^2, IV, day 1 of Q3W
Drug: Docetaxel — Docetaxel 75 mg/m^2, IV, day 1 of Q3W
Drug: Liposomal paclitaxel — Liposomal paclitaxel 135-175 mg/m^2, IV, day 1 of Q3W
Drug: Fluorouracil — Fluorouracil 750 mg/m^2, IV, day 1-5 of Q3W

SUMMARY:
This study is a prospective, open-label, multi-center phase III study; patients with untreated stage IIIA to stage IVB head and neck squamous cell carcinoma (including oral cavity cancer, oropharyngeal cancer, hypopharyngeal cancer, and laryngeal cancer) who meet the inclusion criteria are randomized 1:1 and given pembrolizumab 200 mg d1+ chemotherapy for 2 cycles (experimental group), 2 cycles of chemotherapy (control group), and then stratified according to the patient's condition. If the imaging evaluation after neoadjuvant treatment is (complete response, CR), adjuvant radiotherapy will be given; if the imaging evaluation is (partial response, PR) or (stable disease, SD), surgery (within 2 weeks) will be performed, followed by standard treatment. The main research hypothesis of this study: pembrolizumab combined with standard chemotherapy can significantly improve the rate of pathological complete response (pCR) compared with standard chemotherapy.

DETAILED DESCRIPTION:
This study is a prospective, open-label, multi-center phase III study; Patients with untreated stage IIIA to stage IVB head and neck squamous cell carcinoma (including oral cavity cancer, oropharyngeal cancer, hypopharyngeal cancer, and laryngeal cancer) who met the inclusion criteria were randomized in a 1:1 ratio and given 2 cycles of pembrolizumab 200 mg d1 + chemotherapy (see the table below for detailed chemotherapy regimens) (experimental group) and 2 cycles of chemotherapy (control group), and were divided according to the patient's condition. layer. If the imaging evaluation is CR after neoadjuvant treatment, radiotherapy (60-70Gy) ± chemotherapy (investigator's choice) will be given as adjuvant treatment; if the imaging evaluation is PR or SD, surgery (within 2 weeks) will be performed, and then standard treatment will be given. treat. If the imaging evaluation is PD, standard treatment will be given. Enrolled patients must closely monitor the adverse reactions of chemotherapy and record the time, grade, treatment measures, outcomes, etc. All patients were reviewed every 3 months for 1 year; after 1 year, they were reviewed every 6 months for 3 years; patient recurrence and survival data were recorded.

The investigators speculate that, compared with the traditional induction chemotherapy regimen, the induction chemotherapy regimen of pembrolizumab combined with chemotherapy may be safer and more effective, and easier for clinical application. At present, there are no research reports on the induction chemotherapy of pembrolizumab combined with cisplatin and nab-paclitaxel for patients with locally advanced operable head and neck squamous cell carcinoma. We intend to conduct a randomized controlled study on the efficacy and safety of pembrolizumab combined with chemotherapy as neoadjuvant therapy in Chinese patients with operable head and neck squamous cell carcinoma, and provide a basis for the neoadjuvant therapy of pembrolizumab combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage IIIA-IVB head and neck squamous cell carcinoma confirmed by histology and/or cytology;
2. Have not received immunotherapy in the past;
3. The researchers believe that he can safely receive pembrolizumab combined with chemotherapy or neoadjuvant chemotherapy;
4. Age ≥18 years;
5. ECOG 0-2;
6. Measurable disease as defined by RECIST v1.1;
7. Organs function normally;
8. Female and male participants of reproductive potential must agree to use appropriate contraception throughout the study period and for 180 days after the last study treatment;
9. Male participants must not donate sperm throughout the study and for 180 days after the last study treatment.

Exclusion Criteria:

1. Presence of distant metastasis;
2. Female subjects with a positive urine pregnancy test within 72 hours before the start of the study or within 24 hours after starting radiation therapy (with or without cisplatin);
3. received a live vaccine within 30 days before enrollment;
4. Diagnosed with immunodeficiency or receiving systemic steroid treatment or any other form of immunosuppressive treatment within 7 days before enrollment;
5. Have imaging detectable (even if asymptomatic and/or previously treated) central nervous system metastases and/or cancerous meningitis;
6. Have undergone surgery before commencing the study or have failed to recover adequately from toxicity or complications resulting from the intervention;
7. Previous allogeneic tissue/solid organ transplant;
8. Severe hypersensitivity reaction (≥Grade 3) to pembrolizumab or any of its excipients, radiotherapy, platinum, paclitaxel, 5-FU or their analogs;
9. Have an active autoimmune disease requiring systemic therapy in the past 2 years;
10. History of (non-infectious) pneumonia requiring steroid treatment;
11. Have a history of human immunodeficiency virus (HIV) infection;
12. Have a history of hepatitis B or be positive for hepatitis B virus (defined as a positive reaction to hepatitis B surface antigen [HBsAg]) or active hepatitis C (defined as detection of hepatitis C virus [HCV] ribonucleic acid).
13. Have any medical history, treatment, or laboratory abnormalities that could confound the study results, interfere with participant participation throughout the study, or be detrimental to the best interests of the participant (e.g., Hashimoto's thyroiditis, etc.);
14. Have a known history of mental illness or substance abuse disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) of pembrolizumab combined with standard chemotherapy neoadjuvant therapy in patients with locally advanced head and neck squamous cell carcinoma | 12 week
  pCR was defined as the absence of residual invasive squamous cell carcinoma within the primary tumor specimen on resection/needle biopsy
Pathological complete response rate (pCR) of standard chemotherapy neoadjuvant chemotherapy in patients with locally advanced head and neck squamous cell carcinoma | 12 week
  pCR was defined as the absence of residual invasive squamous cell carcinoma within the primary tumor specimen on resection/needle biopsy

SECONDARY OUTCOMES:
The objective response rate (ORR) of neoadjuvant therapy with pembrolizumab combined with standard chemotherapy | 12 week
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1
The objective response rate (ORR) of neoadjuvant chemotherapy with standard chemotherapy | 6 week
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1
The 1-year and 2-year event-free survival rates (1y-EFS, 2y-EFS) after pembrolizumab combined with standard chemotherapy neoadjuvant therapy | 2 year
  EFS is defined as the time from randomization to any event, including disease progression, discontinuation of treatment for any reason, or death
The 1-year and 2-year event-free survival rate (1y-EFS, 2y-EFS) after neoadjuvant chemotherapy with standard chemotherapy | 2 year
  EFS is defined as the time from randomization to any event, including disease progression, discontinuation of treatment for any reason, or death
The functional preservation rate of pembrolizumab combined with standard chemotherapy | 3 year
  Functional preservation is defined as preserving and repairing the anatomical structure of the larynx, and reconstructing the breathing and pronunciation functions of the larynx, or protecting the appearance of the tongue and physiological functions such as speech, chewing and swallowing
The functional preservation rate of standard chemotherapy | 3 year
  Functional preservation is defined as preserving and repairing the anatomical structure of the larynx, and reconstructing the breathing and pronunciation functions of the larynx, or protecting the appearance of the tongue and physiological functions such as speech, chewing and swallowing
The 2-year overall survival rate (2y-OS) after Neoadjuvant pembrolizumab combined with standard chemotherapy | 2 year
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
The 2-year overall survival rate (2y-OS) after Neoadjuvant Therapy with standard chemotherapy | 2 year
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
Pathological complete response rate (pCR) of pembrolizumab combined with standard chemotherapy as neoadjuvant therapy in patients of locally advanced head and neck squamous cell carcinoma with CPS (combined positive score) ≥1 | 12 week
  pCR was defined as the absence of residual invasive squamous cell carcinoma in the resected primary lesion specimen
Pathological complete response rate (pCR) of pembrolizumab combined with standard chemotherapy as neoadjuvant therapy in patients of locally advanced head and neck squamous cell carcinoma with CPS (combined positive score) <1 | 12 week
  pCR was defined as the absence of residual invasive squamous cell carcinoma in the resected primary lesion specimen
The 2-year event-free survival rates (2y-EFS) after pembrolizumab combined with standard chemotherapy neoadjuvant therapy with CPS (combined positive score) ≥1 | 2 year
  EFS is defined as the time from randomization to any event, including disease
The 2-year event-free survival rates (2y-EFS) after pembrolizumab combined with standard chemotherapy neoadjuvant therapy with CPS (combined positive score) <1 | 2 year
  EFS is defined as the time from randomization to any event, including disease
The 2-year overall survival rate (2y-OS) after Neoadjuvant pembrolizumab combined with standard chemotherapy with CPS(combined positive score) ≥1 | 2 year
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
The 2-year overall survival rate (2y-OS) after Neoadjuvant pembrolizumab combined with standard chemotherapy with CPS(combined positive score) <1 | 2 year
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
Incidence of Treatment-Emergent Adverse Events (TRAEs) of pembrolizumab combined with standard chemotherapy in neoadjuvant therapy | 3 year
  TRAEs include 5 levels, base on Common Terminology Criteria for Adverse Events (CTCAE) is widely accepted as the standard classification and severity grading scale for adverse events in cancer therapy, clinical trials and other oncology settings.
Incidence of Treatment-Emergent Adverse Events (TRAEs) of neoadjuvant chemotherapy with standard chemotherapy | 3 year
  TRAEs include 5 levels, base on Common Terminology Criteria for Adverse Events (CTCAE) is widely accepted as the standard classification and severity grading scale for adverse events in cancer therapy, clinical trials and other oncology settings.
The quality of life of pembrolizumab combined with standard chemotherapy neoadjuvant therapy measured by KPS (Karnofsky performance status) scores | 3 year
  A standard way of measuring the ability of cancer patients to perform ordinary tasks. The KPS scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities.
The quality of life of standard chemotherapy neoadjuvant therapy measured by KPS (Karnofsky performance status) scores | 3 year
  A standard way of measuring the ability of cancer patients to perform ordinary tasks. The KPS scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Huang, Study Chair — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT06102395/Prot_SAP_002.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT06102395/ICF_001.pdf